CLINICAL TRIAL: NCT04734184
Title: Title A Prospective Study on 18F-DCFPyL PET/CT Imaging in Biochemical Recurrence of Prostate Cancer
Brief Title: A Prospective Study on 18F-DCFPyL PET/CT Imaging in Biochemical Recurrence of Prostate Cancer
Acronym: Python
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Curium PET France (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2020-000121-37
Record Dates: First submitted 2021-01-27; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Prostate Cancer Recurrent

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: DCFPyL — Single dose injection

SUMMARY:
PYTHON is designed to establish the efficacy and safety of 18F-DCFPyL in comparison with that of 18F-fluorocholine, in patients with first biochemical recurrence (BCR) after initial definitive therapy (prostatectomy, external beam radiotherapy or brachytherapy) for histopathologically confirmed prostate adenocarcinoma per original diagnosis. PET/CT scans will be each interpreted by three independent masked experts who are not otherwise involved in the trial.

DETAILED DESCRIPTION:
The primary objective is the per-patient detection rate of 18F-DCFPyL in comparison with 18F-Fluorocholine. Secondary objectives include the assessment of the impact on patient treatment management, the per-region detection rate, the sensitivity and specificity on a per-patient and per-region basis, the concordance rate between both tracers, and the safety. The study was initiated in July 2020, and the recruitment of the planned 217 patients has been completed in October 2020. The follow-up phase is ongoing. Typically, as part of the routine care practice, these patients receive appropriate treatment and follow-up. The investigating sites are therefore requested for the period of 7 months after the second tracer injection, to provide any results of subsequent biopsies, imaging studies, clinical findings, PSA measurements, and disease management, if performed in routine practice. Treatment decisions are locally made at the discretion of the referring physician based on all available clinical information, including the non-masked local reports of both PET/CT and any other imaging results. After completion of the study, a consensus will be obtained from a multidisciplinary independent board (truth panel), based on the surrogate standard of reference which will include all the above-mentioned available results. Assessments will be made on a per-region and per-patient basis. The truth panel will consist in 3 independent experts not otherwise involved in the trial. All above information will be sequentially presented to the truth panel experts. The order of presentation of 18F-FCH PET/CT and 18F-DCFPyl PET/CT results will be randomized. The truth panel will have to assess the impact of each PET/CT examination on disease restaging and change in treatment intent, by filling in a patient management questionnaire after review of each PET/CT examination report.

ELIGIBILITY:
Inclusion Criteria:

1. Male.
2. Age min 18 years.
3. Histopathological proven prostate adenocarcinoma per original diagnosis.
4. First suspected recurrence of prostate cancer based on rising prostate-specific antigen (PSA) after initial curative therapy with radical prostatectomy of PSA ≥ 0.2 ng/mL confirmed by a subsequent PSA value of ≥0.2 ng/mL or with radiation therapy (external beam or brachytherapy) of PSA > 2 ng/mL above the nadir after therapy regardless of the serum concentration of the nadir.
5. Able and willing to provide informed consent and comply with protocol requirements
6. Patient who can undergo all study procedures per Investigator's point of view
7. Patient with social insurance cover.

Exclusion Criteria:

Patients displaying any of the following criteria will not be included:

1. ECOG > 2
2. History of previous salvage therapies (including salvage radiotherapy or salvage lymph node dissection)
3. History of adjuvant radiotherapy
4. History of cryotherapy, high-intensity focused ultrasound (HIFU)
5. Other active malignant tumour
6. Treatment with Androgen Deprivation Therapy (ADT) in the past 30 days or ongoing
7. Treatment with colchicine in the past 8 days or ongoing
8. Treatment with hematopoietic colony stimulating factors (CSF) in the past 5 days or ongoing
9. Unable to lie supine for imaging
10. Known allergy to investigational or reference products or to any excipients
11. Unable to provide written consent (linguistic or psychological inability)
12. Participation in another clinical study within one month prior to inclusion
13. Uncooperative, in the Investigator's opinion.
14. Subjects deprived of their freedom by administrative or legal decision or who are under guardianship

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
to compare per-patient detection rate of 18F-DCFPyL PET/CT versus that of 18F-FCH PET/CT. | 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- CURIUM PET France, Saint-Beauzire, France

IPD SHARING:
Plan to Share IPD: Undecided